CLINICAL TRIAL: NCT04078659
Title: Controlled Hypotension During Endoscopic Sinus Surgery: A Comparison of Propofol and Magnesium Sulfate
Brief Title: Propofol and Magnesium Sulfate Intravenous Infusion During Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS ∕18.08.247
Record Dates: First submitted 2019-08-02; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Endoscopic Sinus Surgery
MeSH Terms: interventions — Lidocaine; Fentanyl; Propofol; Atracurium; Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol infusion (Experimental): Patients received intravenous Propofol infusion
  Interventions: Drug: Propofol infusion; Drug: Lidocaine; Drug: Fentanyl; Drug: Propofol; Drug: Atracurium; Procedure: Mechanical Ventilation
- Magnesium Sulfate infusion (Experimental): Patients received intravenous Magnesium Sulfate infusion
  Interventions: Drug: Magnesium Sulfate infusion; Drug: Lidocaine; Drug: Fentanyl; Drug: Propofol; Drug: Atracurium; Procedure: Mechanical Ventilation

INTERVENTIONS:
Drug: Propofol infusion — Following induction of anaesthesia, propofol infusion will be started 75 mcg/kg/min for the first 10-15 minutes, then a maintenance infusion of propofol (50 mcg/kg /min)
  Arms: Propofol infusion
Drug: Magnesium Sulfate infusion — Before induction of anaesthesia, Magnesium Sulfate infusion will be started at 40 mg/kg in 100 ml saline over 10 minutes as the loading dose then Magnesium sulfate infusion 10-15 mg/kg/hr started immediately after induction of anaesthesia
  Arms: Magnesium Sulfate infusion
Drug: Lidocaine — Patients will receive iv lidocaine 1.5 mg/kg before induction of anaesthesia
Drug: Fentanyl — Patients will receive fentanyl 1-2 mcg/kg before induction of anaesthesia
Drug: Propofol — Patients will receive propofol in a dose of 1-2 mg /kg
Drug: Atracurium — Patients will receive 0.6 mg /kg iv atracurium over 60 sec, to facilitate tracheal intubation
Procedure: Mechanical Ventilation — Patients lungs will be ventilated using the volume controlled mechanically ventilated with 40% oxygen in the air with positive end-expiratory pressure (PEEP) of 5 cmH2O, tidal volume 500 ml and Respiratory Rate of 12 per minute

SUMMARY:
Endoscopic Sinus surgery usually associated by bleeding, despite using of local vasopressor injection, head up position- controlled hypotension is generally used for control of this purpose.

Propofol has been reported as a good agent for controlled hypotension by decreasing systemic vascular resistance secondary to arterial and venous vasodilation and a decrease in myocardial contractility with a dose-dependent property.

Magnesium Sulfate also has been reported as an agent of hypotensive anaesthesia by inhibition of the release of norepinephrine by blocking N-type calcium channel at the nerve ending beside acting as a vasodilator.

The well known pharmacodynamic effects of the intravenous infusion of propofol or Magnesium Sulfate may prove the advantage of this group in controlling intraoperative blood pressure thus reducing surgical field bleeding.

DETAILED DESCRIPTION:
The aim of the work to compare the efficacy of propofol and magnesium sulfate to control blood pressure during endoscopic sinus surgery and the resultant effects on the quality of the surgical field including bleeding and visibility.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Classes I or II

Exclusion Criteria:

* Patients refusal
* Patients with hypersensitivity for any drug used in the study including magnesium, propofol or isoflurane
* Patients receiving magnesium sulfate supplementation
* Patients receiving drugs known to have significant interaction.
* Patients with ischemic heart disease
* Patients with heart defects
* Patients with significant heart failure
* Patients with increased intracranial pressure.
* Patients with systemic hypertension

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Mean arterial blood pressure (MAP) | 15 minutes after the induction of the hypotensive agent
  automatically non invasive measured every 3 minutes , recorded every 15 minutes till the end and 15 minutes after extubation the end and 15 minutes after extubation

SECONDARY OUTCOMES:
The blood loss | at the end of the surgery
  The blood loss would be calculated using the following formula Blood Loss = Blood Volume. In )Hct 1 / Hct2)
The number of patients will need nitroglycerine and dose | at the end of the surgery
  The number of patients will need nitroglycerine
Use of Ephedrine | at the end of the surgery
  The number of patients will need ephedrine
Need for blood transfusion | at the end of the surgery
  The number of patient need for blood transfusion
Postoperative Ramsey sedation | for the first hour postoperative
  patient awake, anxious, agitated or restless 2 patient awake -1co operative, oriented and tranquil 3 patient drowsy with respond to command 4 patient asleep brisk response to glabella tap or loud auditory sound 5 patient asleep with sluggish response to stimulus 6 patient hasno response to nail bed pressure or othernoxious stimuli
Simplified post operative nausea and vomiting score | for the first 24 hour postoperative
  using impact scale score evaluation
Recovery time | one hour after extubation
  time needed to reach modified aldrete score> or=9)
Heart rate (HR) | 15 minutes after the start of the hypotensive agent
surgical field assessment | 2 hours intraoperative
  By the surgeon interms of bleeding and visibility using a 6-option Liker-scale scale adapted from Fromme el al. (26): 0 = no bleeding; 1 = minor bleeding, but no aspiration required; 2 = minor bleeding, aspiration required; 3 = minor bleeding, frequent aspiration required; 4 = moderate bleeding, visible� only with aspiration; 5 = severe bleeding, continuous aspiration required

CONTACTS AND LOCATIONS:
Overall Officials: Hazem E Moawed, Study Director — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Nabil A Abd El-Mageed, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes